CLINICAL TRIAL: NCT05736822
Title: The Impact of the COVID-19 Pandemic on the Patient in Need of an Intervention - COVID Surg III
Brief Title: The Impact of the COVID-19 Pandemic on the Patient in Need of an Intervention
Acronym: COVID Surg III
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 15813
Record Dates: First submitted 2023-02-20; First posted 2023-02-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Surgical Procedures, Operative; COVID-19; SARS-CoV-2
Keywords: Specialties, Surgical; Surgery Department, Hospital
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mixed-method observational study: the impact of pandemic related changes in healthcare on quality of life and experiences with healthcare in Dutch patients undergoing surgery or another intervention during the covid pandemic (2020-2021).

Phase 1: qualitative study to gain insight in relevant themes in Patient Reported Experiences Measures (PREMs) by conducting focus groups Phase 2: creating and validating a questionnaire based on themes identified in phase 1 Phase 3: questionnaire study among Dutch patients who underwent an intervention in 2020-2021 using the validated questionnaire of phase 2. The answers will be linked to data from national patients registries in surgery, cardiology, orthopedics and neurology.

ELIGIBILITY:
Inclusion Criteria:

* undergoing surgery or intervention in the Netherlands in 2020 or 2021

Exclusion Criteria:

* participation language restricted to Dutch

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: (former) surgical, orthopedic, cardiological patients
Sampling Method: Non-Probability Sample
Enrollment: 5277 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Patient Reported Experience Measures | 2020-2021
  [will be specified based on phase 1 of the study, see description]

CONTACTS AND LOCATIONS:
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD; the available dataset is anonymised and cannot be linked to other datasets.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: from 01-01-2027 until 30-04-2039
Access Criteria: The anonymised dataset is available upon request to the principal investigator Prof. Schelto Kruijff. Requests can be send by email and should include a description of the study objective, primary and secondary outcomes, other data sources that will be used (if applicable), and a brief analysis plan. After discussion within the COVID Surg III research collective, the PI will decide whether or not the dataset will be shared with the requesting researcher. After a positive decision a data sharing agreement will be drafted and signed before the data is shared via a secured digital pathway, for example Zivver.